CLINICAL TRIAL: NCT01760135
Title: Nutritional Requirement for the Severe Trauma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, Director, Surgical Intensive Care Unit, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-001
Record Dates: First submitted 2012-12-21; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Trauma
Keywords: trauma; nutrition; hyperglycemia
MeSH Terms: conditions — Wounds and Injuries; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low calory (Experimental): 15kcal/kg caloric supplement
  Interventions: Dietary Supplement: high caloric nutritional supplement
- high calory (Active Comparator): 25kcal/kg
  Interventions: Dietary Supplement: low caloric nutritional supplement

INTERVENTIONS:
Dietary Supplement: high caloric nutritional supplement — high caloric nutritional supplement (25kcal/kg)
  Arms: low calory
Dietary Supplement: low caloric nutritional supplement — low caloric nutritional supplement(15kcal/kg)
  Arms: high calory

SUMMARY:
After severe trauma, high caloric nutrition supplement do harm on metabolic and immunologic aspects.

ELIGIBILITY:
Inclusion Criteria:

* ISS more than 15 score
* older than 20 years old
* patient who need parenteral nutrition more than 5 days

Exclusion Criteria:

* patients who have metabolic disease except for diabetes
* patients who cannot resuscitated
* very low body weight (< 40kg)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotics usage (days) | participants will be followed for the duration of hospital stay, an expected average of 2 week).

SECONDARY OUTCOMES:
Mortality | participants will be followed for the duration of hospital stay, an expected average of 2 week
Number of date when is showing hyperglycemia (more than 200mg/dL) | participants will be followed for the duration of hospital stay, an expected average of 2 week
Hospitals stays | participants will be followed for the duration of hospital stay, an expected average of 2 week
ICU stays | participants will be followed for the duration of hospital stay, an expected average of 2 week

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Kyung Hong, MD, PhD., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea